CLINICAL TRIAL: NCT05015231
Title: Multiparametric MRI for Assessment of Changes of Renal Hemodynamics After Fistula Closure in Kidney Transplant Patients: a Pilot Study
Brief Title: Multiparametric MRI for Assessment of Changes of Renal Hemodynamics After Fistula Closure in Kidney Transplant Patients
Acronym: FISCLO
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-00474
Record Dates: First submitted 2021-08-09; First posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Echocardiography; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Echocardiography and MRI — Echocardiography and renal MRI before and after fistula closure

SUMMARY:
Assessment of changes of renal hemodynamics by multiparametric MRI after closure of AVF access.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age > 18 years
* Patients wishing to close the fistula and planned for surgical fistula closure
* eGFR CKD EPI ≥ 45 ml/min/1.73m2 at one year post transplantation
* Stable eGFR within the past 6 months
* Controlled blood pressure

Exclusion Criteria:

* Kidney Transplantation < 12 months before fistula closure
* Proteinuria > 500mg/d
* Presence of donor specific antibodies
* Rejection within the past 6 months
* BK virus replication within the past 3 months
* Cardiac pacemaker, which is not compatible with MRI
* Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients with a functioning graft and a patent hemodialysis fistula
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of changes in renal hemodynamics by multiparametric MRI after closure of AVF access | evaluation of short term changes within 2 weeks after fistula closure and longterm changes 6 months after fistula closure
  Assessing changes in renal perfusion
Assessment of changes in renal hemodynamics by multiparametric MRI after closure of AVF access | evaluation of short term changes within 2 weeks after fistula closure and longterm changes 6 months after fistula closure
  Assessing changes in renal oxygenation

SECONDARY OUTCOMES:
Correlation between AVF access flow and changes as assessed during pneumatic fistula compression with changes in renal hemodynamics after fistula closure | evaluation of short term changes within 2 weeks after fistula closure and longterm changes 6 months after fistula closure
  Correlation between AVF access flow and changes as assessed during pneumatic fistula compression with changes in renal hemodynamics after fistula closure

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Müller, Professor, Principal Investigator — University Hospital Zurich, Nephrology
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No